CLINICAL TRIAL: NCT05637931
Title: Evaluation of Circulating PlexinD1 as a Potential Biomarker of Polymyositis and Dermatomyositis.
Brief Title: Plexin D1 as a Potential Biomarker inPM/DM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Khalifa Ali Khalifa, doctor, Assiut University
Other Study IDs: plexinD1 in PM/DM
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Polymyositis; Dermatomyositis
MeSH Terms: conditions — Polymyositis; Dermatomyositis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- adult polymyositis and dermatomyositis
  Interventions: Diagnostic Test: plexinD1
- juvenile dermatomyositis
  Interventions: Diagnostic Test: plexinD1
- healthy controls
  Interventions: Diagnostic Test: plexinD1

INTERVENTIONS:
Diagnostic Test: plexinD1 — evaluation of the serum level of plexinD1

SUMMARY:
evaluation of level of serum circulating plexin D1 on extacellular vesicles in adult PM/DM patients and juvenile dermatomysitis.

DETAILED DESCRIPTION:
Polymyositis (PM) and dermatomyositis (DM) are autoimmune inflammatory diseases that primarily target muscle.

autoimmune Dermatomyositis (DM) is a rare inflammatory disease that mainly affects skin, muscle, and lung.

Inflammatory myopathies (IMs) often have distinct histopathologic features suggesting humorally mediated involvement of the microcirculation in dermatomyositis (DM), including early capillary deposition of the complement C5b-9 membranolytic attack complex (MAC) and secondary ischaemic changes; and CD8 T-cell-mediated and MHC1-restricted autoimmune attack of myofibers in polymyositis (PM) and inclusion body myositis.

Plexins are a conserved family of large proteins (~200kDa) that are the canonical receptors for semaphorin molecules. Plexins are divided into four classes, A through D.

Recently, plexin and semaphorin molecules have been shown to control cell movement and cell-cell interaction in the immune system .

Extracellular vesicles (EVs) are lipid bilayer membrane vesicles that exist in various bodily fluids. EVs are released by normal, diseased, and transformed cells in vitro and in vivo and are capable of carrying lipids, proteins, mRNAs, non-coding RNAs, and even DNA. They are abundant in serum and plasma and have been a source of considerable interest as potential disease biomarkers. Normally, they maintain physiological functions by transferring biological information to neighboring cells and facilitating intercellular communication, but are also involved in the pathogenesis of numerous autoimmune diseases LC/MS analysis identified 1220 proteins in serum EVs. Of these, plexin D1 was enriched in those from PM/DM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult PM/DM patients .
2. Juvenile dermatomyositis patients.

Exclusion Criteria:

* 1-Patients with other autoimmune diseases ( rheumatoid arthritis ,systemic lupus erythematosus, polyarteritis nodosa sarcoidosis, scleroderma, spondylarthritis and inflammatory bowel disease) 2-Patients with malignant tumors 3-Patients with active infection 4-Patients with severe heart, lung, and kidney dysfunction

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 3 groups under the study adult polymyositis and dermatomyositis,juvenile dermatomyositis. and healthy control .22 subjects in each group.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2022-12-25 (Estimated); Primary Completion 2023-12-25 (Estimated); Study Completion 2024-01-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of circulating PlexinD1 as a potential biomarker of polymyositis and dermatomyositis. | baseline
  evaluation of plexinD1in PM/DM patients

CONTACTS AND LOCATIONS:
Overall Officials: Eman Ahmed Hamed Omran, professor, Study Director — Assiut University; Manal Hassanien, professor, Study Director — Assiut University; Ahmed Abdel Khalek Hafez, lecturer, Study Director — Assiut University; Helal F. Hetta, professor, Study Director — Assiut University

REFERENCES:
- [Background] Ytterberg SR. Treatment of refractory polymyositis and dermatomyositis. Curr Rheumatol Rep. 2006 Jun;8(3):167-73. doi: 10.1007/s11926-996-0021-7. PMID 16901073
- [Background] Li Y, Bax C, Patel J, Vazquez T, Ravishankar A, Bashir MM, Grinnell M, Diaz D, Werth VP. Plasma-derived DNA containing-extracellular vesicles induce STING-mediated proinflammatory responses in dermatomyositis. Theranostics. 2021 May 21;11(15):7144-7158. doi: 10.7150/thno.59152. eCollection 2021. PMID 34158841
- [Background] Feldman BM, Rider LG, Reed AM, Pachman LM. Juvenile dermatomyositis and other idiopathic inflammatory myopathies of childhood. Lancet. 2008 Jun 28;371(9631):2201-12. doi: 10.1016/S0140-6736(08)60955-1. PMID 18586175
- [Background] Gherardi RK. Pathogenic aspects of dermatomyositis, polymyositis and overlap myositis. Presse Med. 2011 Apr;40(4 Pt 2):e209-18. doi: 10.1016/j.lpm.2010.12.013. Epub 2011 Mar 3. PMID 21376512
- [Background] Devhare PB, Ray RB. Extracellular vesicles: Novel mediator for cell to cell communications in liver pathogenesis. Mol Aspects Med. 2018 Apr;60:115-122. doi: 10.1016/j.mam.2017.11.001. Epub 2017 Nov 11. PMID 29122679
- [Background] Lane RE, Korbie D, Hill MM, Trau M. Extracellular vesicles as circulating cancer biomarkers: opportunities and challenges. Clin Transl Med. 2018 May 31;7(1):14. doi: 10.1186/s40169-018-0192-7. PMID 29855735
- [Background] Turpin D, Truchetet ME, Faustin B, Augusto JF, Contin-Bordes C, Brisson A, Blanco P, Duffau P. Role of extracellular vesicles in autoimmune diseases. Autoimmun Rev. 2016 Feb;15(2):174-83. doi: 10.1016/j.autrev.2015.11.004. Epub 2015 Nov 7. PMID 26554931
- [Background] Uto K, Ueda K, Okano T, Akashi K, Takahashi S, Nakamachi Y, Imanishi T, Awano H, Morinobu A, Kawano S, Saegusa J. Identification of plexin D1 on circulating extracellular vesicles as a potential biomarker of polymyositis and dermatomyositis. Rheumatology (Oxford). 2022 Apr 11;61(4):1669-1679. doi: 10.1093/rheumatology/keab588. PMID 34297034